CLINICAL TRIAL: NCT04988867
Title: An Open-Label Study of Trofinetide for the Treatment of Girls Two to Five Years of Age Who Have Rett Syndrome
Acronym: DAFFODIL™
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: As a result of marketing approval of trofinetide on 10 March 2023, the study was terminated by the Sponsor with the intent of switching patients to commercially available product.
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-2566-009
Record Dates: First submitted 2021-07-23; First posted 2021-08-04 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — trofinetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - trofinetide (Experimental): Oral dose of trofinetide
  Interventions: Drug: Trofinetide

INTERVENTIONS:
Drug: Trofinetide — Trofinetide solution of 10-30 mL based on subject's weight at Baseline, administered twice daily by mouth or gastrostomy tube (G-tube)

SUMMARY:
To investigate the safety and tolerability of long-term treatment with oral trofinetide in girls with Rett syndrome

ELIGIBILITY:
Inclusion Criteria:

* Female subject

  1. 2 to 4 years of age and body weight ≥9 kg and <20 kg at Screening OR
  2. 5 years of age and body weight ≥9 kg and <12 kg at Screening
* Can swallow the study medication provided as a liquid solution or can take it by gastrostomy tube
* The subject's caregiver is English-speaking and has sufficient language skills to complete the caregiver assessments
* Has classic/typical Rett syndrome (RTT) or possible RTT according to the Rett Syndrome Diagnostic Criteria
* Has a documented disease-causing mutation in the MECP2 gene
* Has a stable pattern of seizures, or has had no seizures, within 8 weeks prior to Screening
* Subject and caregiver(s) must reside at a location to which study drug can be delivered and have been at their present residence for at least 4 weeks prior to Screening

Exclusion Criteria:

* Has been treated with insulin within 12 weeks of Baseline
* Has current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, Type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus), renal, hepatic, respiratory or gastrointestinal disease (such as celiac disease or inflammatory bowel disease) or has major surgery planned during the study
* Has a history of, or current, cerebrovascular disease or brain trauma
* Has significant, uncorrected visual or uncorrected hearing impairment
* Has a history of, or current, malignancy
* Has any of the following:

  1. QTcF interval of >450 ms at Screening or Baseline
  2. History of a risk factor for torsades de pointes (e.g., heart failure or family history of long QT syndrome)
  3. History of clinically significant QT prolongation that is deemed to put the subject at increased risk of clinically significant QT prolongation
  4. Other clinically significant finding on ECG at Screening or Baseline

Additional inclusion/exclusion criteria apply. Patients will be evaluated at baseline to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all prespecified entry criteria).

Ages: 2 Years to 5 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Colorado, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital/Harvard Medical School, Boston, Massachusetts
  - Gillette Children's Hospital, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Percy AK, Ryther R, Marsh ED, Neul JL, Benke TA, Berry-Kravis EM, Feyma T, Lieberman DN, Ananth AL, Fu C, Buhrfiend C, Barrett A, Doshi D, Darwish M, An D, Bishop KM, Youakim JM. Results from the phase 2/3 DAFFODIL study of trofinetide in girls aged 2-4 years with Rett syndrome. Med. 2025 Jun 13;6(6):100608. doi: 10.1016/j.medj.2025.100608. Epub 2025 Mar 4. PMID 40043705
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385

RESULTS

PARTICIPANT FLOW:
Groups:
- Trofinetide: Trofinetide oral solution was administered twice daily for up to approximately 26 months, orally or administered by gastrostomy (G) tube.
Period: Overall Study
Arm/Group | Trofinetide
Started | 15
Completed | 0
Not Completed | 15
Not completed — Study terminated by Sponsor | 12
Not completed — Adverse Event | 2
Not completed — Study drug noncompliance | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled and treated
Arm/Group | Trofinetide
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Treatment With Oral Trofinetide
Description: Percentage of patients with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), withdrawals due to AEs, potentially clinically important (PCI) changes in other safety assessments (laboratory values, vital signs, or ECGs, following protocol-defined PCI criteria)
Time Frame: Mean study drug exposure 434 days, corresponding to 1.2 years
Population: All patients enrolled and treated
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 15
Participants
  Patients with TEAEs | 14
  Patients with SAEs | 4
  Patients with AEs leading to discontinuation | 2
  Alanine transaminase ≥3 ULN | 1
  Aspartate transaminase ≥3 ULN | 1
  Potassium ≤3.0 mmol/L | 1
  Leukocytes ≥15 × 10Ê9/L | 2
  Neutrophils ≤1.5 × 10E9/L | 2
  Hematocrit <0.3 | 1
  Hemoglobin <100 g/L | 1

2. Primary Outcome: AUC0-12,ss (Area Under the Concentration-time Curve From Time 0 to 12 h at Steady State)
Description: Area under the concentration-time curve from time 0 to 12 h at steady state as obtained from population pharmacokinetic (PK) modelling
Time Frame: PK samples were taken predose and at Weeks 2, 4, 8, and 12
Population: Patients enrolled, treated, and with at least one quantifiable PK concentration
Measure: Mean (Standard Deviation); unit: μg x h/mL
Arm/Group | Trofinetide
Number analyzed (Participants) | 13
μg x h/mL | 1015.7 (135.9)

3. Primary Outcome: Cmax,ss (Maximum Observed Drug Concentration at Steady State)
Description: Maximum observed drug concentration at steady state as obtained from population pharmacokinetic (PK) modelling
Time Frame: PK samples were taken predose and at Weeks 2, 4, 8, and 12
Population: Patients enrolled, treated, and with at least one quantifiable PK concentration
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Trofinetide
Number analyzed (Participants) | 13
μg/mL | 181.5 (22.8)

4. Primary Outcome: Cmin,ss (Minimum Observed Drug Concentration at Steady State of Oral Trofinetide)
Description: Minimum observed drug concentration at steady state of oral trofinetide as obtained from population pharmacokinetic (PK) modeling
Time Frame: PK samples were taken predose and at Weeks 2, 4, 8, and 12
Population: Patients enrolled, treated, and with at least one quantifiable PK concentration
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Trofinetide
Number analyzed (Participants) | 13
μg/mL | 19.6 (6.3)

5. Primary Outcome: Tmax (Time of the Maximum Observed Drug Concentration at Steady State)
Description: Time of the maximum observed drug concentration at steady state as obtained from population pharmacokinetic (PK) modelling
Time Frame: PK samples were taken predose and at Weeks 2, 4, 8, and 12
Population: Patients enrolled, treated, and with at least one quantifiable PK concentration
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Trofinetide
Number analyzed (Participants) | 13
h | 1.8 (0.2)

ADVERSE EVENTS:
Time Frame: Mean study drug exposure 434 days, corresponding to 1.2 years
Arm/Group | Trofinetide
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=15)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroenteritis sapovirus (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Rett syndrome (Congenital, familial and genetic disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (26)
Vomiting (Gastrointestinal disorders) | 8 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
COVID-19 (Infections and infestations) | 7 (9)
Gastroenteritis (Infections and infestations) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (7)
Influenza (Infections and infestations) | 3 (3)
Conjunctivitis (Infections and infestations) | 2 (3)
Ear infection (Infections and infestations) | 2 (3)
Candida infection (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (2)
Otitis media acute (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 5 (9)
Epilepsy (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (2)
Irritability (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As a result of marketing approval of trofinetide on 10 March 2023, the study was terminated by the Sponsor with the intent of switching patients to commercially available product. The study was terminated on 31 May 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04988867/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04988867/SAP_001.pdf